CLINICAL TRIAL: NCT03305809
Title: Effect of LY3154207 on Cognition in Mild-to-Moderate Dementia Due to Lewy Body Dementia (LBD) Associated With Idiopathic Parkinson's Disease (PD) or Dementia With Lewy Bodies (DLB)
Brief Title: A Study of LY3154207 in Participants With Dementia Due to Lewy Body Dementia (LBD) Associated With Idiopathic Parkinson's Disease (PD) or Dementia With Lewy Bodies (DLB)
Acronym: PRESENCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16261; I7S-MC-HBEH (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-10-04; First posted 2017-10-10 (Actual); Results first posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Lewy Body Dementia
Keywords: Parkinson Disease Dementia; Parkinson Disease; Dopamine; Cognition; Lewy Body Dementia; Dementia with Lewy Bodies
MeSH Terms: conditions — Lewy Body Disease; Parkinson Disease | interventions — LY3154207

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo administered orally once a day (QD).
  Interventions: Drug: Placebo
- 10 milligram (mg) LY3154207 (Experimental): Participants received 10 mg LY3154207 administered orally QD.
  Interventions: Drug: LY3154207
- 30 mg LY3154207 (Experimental): Participants received 30 mg LY3154207 administered orally QD.
  Interventions: Drug: LY3154207
- 75 mg LY3154207 (Experimental): Participants received 75 mg LY3154207 administered orally QD.
  Interventions: Drug: LY3154207

INTERVENTIONS:
Drug: LY3154207 — Administered orally.
  Arms: 10 milligram (mg) LY3154207; 30 mg LY3154207; 75 mg LY3154207
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
A randomized placebo-controlled trial to evaluate the safety and efficacy of three doses of study drug LY3154207 treated for 12 weeks in participants with mild-to-moderate dementia associated with LBD (PDD or DLB).

ELIGIBILITY:
Inclusion Criteria:

* Have dementia as defined by a decline in cognitive function, which in the opinion of the investigator has resulted in functional impairment.
* Meet diagnostic criteria for PD per MDS criteria or DLB per 4th Consensus Report of the DLB Consortium.
* Have a score on the MoCA of 10 - 23.
* Are Modified Hoehn and Yahr Stages 0 - 4.
* Have a blood pressure (BP) or pulse rate at screening and randomization, as determined by three sequential BP/pulse rate measurements in a seated position:

  * Participants <60 years old:

    1. A mean systolic BP less than or equal to 140 millimeters of mercury (mmHg), a mean diastolic BP less than or equal to 90 mmHg and a mean pulse rate less than or equal 90 beats/minute in a seated position.
    2. Each of the 3 systolic BP measurement must be less than 180 mmHg
  * Participants ≥60 years old:

    1. A mean systolic BP less than or equal to 150 mmHg, a mean diastolic BP less than or equal to 90 mmHg and a mean pulse rate less than or equal to 90 beats/min in a seated position.
    2. Each of the 3 systolic BP measurement must be less than 180 mmHg
* If on anti-parkinsonian agents, participants must be on stable dosage for at least 3 weeks prior to screening, and should remain on stable doses during the course of the study.
* If on medications affecting cognition (rivastigmine, galantamine, donepezil, memantine), participants must be on stable dosage for at least 3 weeks prior to screening and should remain at a stable dosage during the course of the study.
* If on antidepressant medications, participants must be on stable dosage for at least 3 weeks prior to screening and should remain at a stable dosage during the course of the study.
* If on clozapine, quetiapine, and pimavanserin to address drug induced or disease related psychosis, participants must be on stable dosage for 3 weeks prior to screening and should remain at a stable dosage during the course of the study.
* If on antihypertensive medications, participants must be on stable dosage for at least 3 weeks prior to screening.
* Men should use appropriate contraception.
* All participants must have a reliable caregiver who is in frequent contact with the participant (defined as at least 10 hours per week) and will accompany the participant to screening, baseline, day 7, day 42, day 84 and follow-up.

Exclusion Criteria:

* Are women of childbearing potential.
* Have significant central nervous system or psychiatric disease, other than PD or DLB, that in the investigator's opinion may affect cognition or the ability to complete the study.
* Have a history in the last 6 months of transient ischemic attacks or ischemic stroke.
* Have a history of intra cerebral hemorrhage due to hypertension.
* Have a history of hypertensive encephalopathy.
* Have atypical or secondary parkinsonism due to drugs (e.g., antipsychotics) or disease (such as progressive supranuclear palsy, essential tremor, multiple system atrophy (e.g. striatonigral degeneration, olivopontocerebellar atrophy), or postencephalitic parkinsonism).
* Have a current implantable intracranial stimulator or history of intracranial ablation surgery (e.g., subthalamic, globus pallidus-internal segment [GPi]).
* Have a history of substance abuse within the past 1 year (drug categories defined by the Diagnostic and Statistical Manual of Mental Disorder, 5th Edition [DSM-5], and/or substance dependence within the past 1 year, not including caffeine and nicotine.
* Have a serious or unstable medical illness, other than idiopathic LBD (PDD or DLB), including cardiovascular, hepatic, respiratory, hematologic, endocrinologic, neurologic, or renal disease, or clinically significant laboratory or electrocardiogram (ECG) abnormality as determined by the investigator.

  * Have a history in the last 6 months of exertional angina, unstable angina, myocardial infarction, and acute coronary syndrome.
  * Have a history of heart failure of either New York Heart Association Class III or IV.
  * A history of additional risk factors for Torsades de Pointes (TdP; [e.g., chronic hypokalemia, family history of Long QT Syndrome]).
* Participants with acute liver disease (e.g. acute viral hepatitis, alcoholic hepatitis); participants with a known chronic liver disease (e.g. hepatitis B, C, alcoholic liver disease, cirrhosis); alanine aminotransferase (ALT) or aspartate aminotransferase (AST) equal to or higher than 2X upper limit of normal (ULN); total bilirubin (TBL) equal to or higher than 1.5X ULN; (except for participants with Gilbert's syndrome); or alkaline phosphatase (ALP) equal to or higher than 2X ULN.
* Participants have answered 'yes' to either Question 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) or Question 5 (Active Suicidal Ideation with Specific Plan and Intent) on the "Suicidal Ideation" portion of the Columbia Suicide Severity Rating Scale (C-SSRS)- Children's version, or answer "yes" to any of the suicide-related behaviors (actual attempt, interrupted attempt, aborted attempt).
* Have used antipsychotic medications, with the exception of clozapine, quetiapine, pimavanserin in the 6 months prior to screening and at any time during the course of the study.
* Have used anticholinergics trihexyphenidyl and benztropine in the 4 weeks prior to screening and at any time during the course of the study.
* Have motor conditions for which the antiparkinsonian treatment is expected to change during the course of the study, as well as unpredictable motor fluctuations that in the investigator's opinion would interfere with administering assessments.
* Are taking any medications or food, herbal or dietary supplements that are inhibitors (e.g., ketoconazole, grapefruit juice), or strong/moderate inducers of cytochrome P450 3A4 (CYP3A4) (e.g., rifampicin) or are unable or unwilling to discontinue usage of them 4 weeks prior to first dose of study drug.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (77):
- United States (71):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - Mayo Clinic of Scottsdale, Scottsdale, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - University of Arizona Health Sciences, Tucson, Arizona
  - Parkinson'S & Movement Disorder Institute, Fountain Valley, California
  - University of CA, Irvine, Irvine, California
  - Collaborative Neuroscience Network - CNS, Long Beach, California
  - University of Southern California School of Medicine, Los Angeles, California
  - Pacific Neuroscience Medical Group, Oxnard, California
  - Stanford Neuroscience Health Center, Palo Alto, California
  - SC3 Research Group Inc Pasadena, Pasadena, California
  - SC3 Research Group Inc Reseda, Reseda, California
  - University of California, Davis - Health Systems, Sacramento, California
  - University of Colorado Hospital, Aurora, Colorado
  - Denver Neurological Research, Denver, Colorado
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - New England Institute for Clinical Research, Stamford, Connecticut
  - Hartford Healthcare Chase Movement Disorders Center, Vernon, Connecticut
  - Christiana Care Health Service, Newark, Delaware
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - JEM Research Institute, Atlantis, Florida
  - Visionary Investigators Network, Aventura, Florida
  - Parkinson's Disease and Movement Disorders, Boca Raton, Florida
  - Norman Fixel Institute for Neurological Diseases (FIND), Gainesville, Florida
  - ClinCloud, LLC, Maitland, Florida
  - Visionary Investigators Network, Miami, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - VIN - Victor Faradji, Miami, Florida
  - Collier Neurologic Specialists, Naples, Florida
  - Renstar Medical Research, Ocala, Florida
  - Compass Research, Orlando, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Visionary Investigators Network -VIN-Margarita Almeida, Pembroke Pines, Florida
  - Axiom Research, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Atlanta Center of Medical Research, Atlanta, Georgia
  - Central DuPage Hospital, Winfield, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Josephson Wallack Munshower Neurology, Indianapolis, Indiana
  - University of Kansas School of Medicine, Kansas City, Kansas
  - Maine Neurology, Scarborough, Maine
  - New England Neurological Associates, PC, Methuen, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - QUEST Research Institute, Farmington Hills, Michigan
  - Clinical Research Professionals, Chesterfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Cleveland Clinic of Las Vegas, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - The Cognitive and Research Center of NJ, Springfield, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Dent Neurological Institute, Amherst, New York
  - Alzheimer's Disease and Memory Disorders Center, Buffalo, New York
  - Adirondack Medical Research, Glens Falls, New York
  - Parker Jewish Insititue for Heatlh Care and Rehabilition, New Hyde Park, New York
  - NYU Langone, New York, New York
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Penn State Univ. Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Neurology, PA, Dallas, Texas
  - Neurology Consultants of Dallas, PA, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Research Ins, Houston, Texas
  - Sentara Neurology Specialists, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Evergreen Professional Plaza, Kirkland, Washington
  - University of Wisconsin-Madison Hospital and Health Clinic, Madison, Wisconsin
- Canada (2):
  - Toronto Memory Program, Toronto, Ontario
  - Ottawa Hospital Research Institute, Ottawa
- Puerto Rico (4):
  - Cortex, PSC, Las Piedras, PR
  - Instituto de Neurologia Dra. Ivonne Fraga, San Juan, PR
  - University of Puerto Rico, San Juan, PR
  - Santa Cruz Behavioral PSC, Bayamón

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Chen C, Kowahl NR, Rainaldi E, Burq M, Munsie LM, Battioui C, Wang J, Biglan K, Marks WJ Jr, Kapur R. Wrist-worn sensor-based measurements for drug effect detection with small samples in people with Lewy Body Dementia. Parkinsonism Relat Disord. 2023 Apr;109:105355. doi: 10.1016/j.parkreldis.2023.105355. Epub 2023 Mar 4. PMID 36905719
- [Derived] Wilbraham D, Biglan KM, Svensson KA, Tsai M, Kielbasa W. Safety, Tolerability, and Pharmacokinetics of Mevidalen (LY3154207), a Centrally Acting Dopamine D1 Receptor-Positive Allosteric Modulator (D1PAM), in Healthy Subjects. Clin Pharmacol Drug Dev. 2021 Apr;10(4):393-403. doi: 10.1002/cpdd.874. Epub 2020 Oct 7. PMID 33029934
- See also: A Study of LY3154207 in Participants With Dementia Due to Lewy Body Dementia (LBD) Associated With Idiopathic Parkinson's Disease (PD) or Dementia With Lewy Bodies (DLB) (PRESENCE) — https://www.lillytrialguide.com/en-US/studies/parkinson-s-disease-dementia/HBEH#?postal=

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | 10 Milligram (mg) LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Started | 86 | 86 | 85 | 87
Received at Least One Dose of Study Drug | 86 | 86 | 85 | 87
Completed | 79 | 78 | 66 | 60
Not Completed | 7 | 8 | 19 | 27
Not completed — Adverse Event | 2 | 2 | 6 | 6
Not completed — Death | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0
Not completed — Sponsor Decision | 1 | 0 | 1 | 8
Not completed — Physician Decision | 0 | 0 | 2 | 4
Not completed — Progressive Disease | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 2 | 3
Not completed — Withdrawal due to Assessment Committee Decision | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 4 | 5 | 2
Not completed — Withdrawal due to Caregiver Circumstances | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo: Participants received placebo administered orally QD.
- 10 mg LY3154207: Participants received 10 mg LY3154207 administered orally QD.
- Total: Total of all reporting groups
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207 | Total
Number analyzed (Participants) | 86 | 86 | 85 | 87 | 344
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.00 (7.02) | 72.50 (6.70) | 71.90 (7.35) | 73.00 (5.21) | 72.60 (6.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 15 | 15 | 59
  Male | 70 | 73 | 70 | 72 | 285
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 9 | 11 | 33
  Not Hispanic or Latino | 77 | 81 | 76 | 75 | 309
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2
  Asian | 2 | 1 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 2 | 2 | 11
  White | 79 | 81 | 81 | 85 | 326
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 3 | 2 | 3 | 2 | 10
  Puerto Rico | 5 | 2 | 4 | 4 | 15
  United States | 78 | 82 | 78 | 81 | 319

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Continuity of Attention (CoA) Composite Score of the Cognitive Drug Research Computerized Cognition Battery (CDR-CCB)
Description: The CDR-CCB tests is designed to evaluate the effects of novel compounds on the quality of cognitive functioning which includes tests of attention (simple and choice reaction time, digit vigilance), working memory (spatial and numeric) and episodic memory (word recognition, picture recognition). Continuity of attention measures speed and accuracy and is calculated from 3 attentional tasks on the CDR computerized battery tests. For continuity of attention, the score range is -999 to 35. A high score reflects someone able to keep his/her mind on a single task for a prolonged period. A negative change from baseline reflects impairment compared to baseline. Data presented are model-based bayesian posterior mean response rates with 95% credible interval.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug, who had the baseline efficacy assessment and had at least 1 postdose efficacy assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Number analyzed (Participants) | 69 | 74 | 65 | 54
Units on a scale | 1.04 [-0.339 to 2.373] | 0.15 [-1.206 to 1.496] | 0.96 [-0.448 to 2.362] | 0.26 [-1.310 to 1.801]
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY3154207; Test type: Superiority; Posterior Mean Difference = -0.89, 95% CI 2-sided [-2.776 to 0.969] — Analyses were conducted using a bayesian mixed-model repeated measures (MMRM), and posterior mean change difference is reported
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY3154207; Test type: Superiority; Posterior Mean Difference = -0.08, 95% CI 2-sided [-1.996 to 1.879] — Analyses were conducted using a bayesian MMRM, and posterior mean change difference is reported
Statistical Analysis 3: Comparison: Placebo vs 75 mg LY3154207; Test type: Superiority; Posterior Mean Difference = -0.78, 95% CI 2-sided [-2.873 to 1.277] — Analyses were conducted using a bayesian MMRM, and posterior mean change difference is reported

2. Secondary Outcome: Change From Baseline on the Alzheimer's Disease Cooperative Study-Clinician Global Impression of Change (ADCS-CGIC) Score
Description: The ADCS-CGIC is a validated categorical measure of change in a participant's clinical condition between baseline and follow-up visits; it is used to assess global clinical status. The ADCS CGIC score is based on direct examination of the participant and an interview of the caregiver. The rater should refer to the baseline ADCS-CGIC worksheets in making a rating. A skilled and experienced clinician who is blinded to treatment assignment rates the participant on a 7-point Likert scale, ranging from 1 (marked improvement) to 7 (marked worsening). 1= Very much better 2= Much better 3= A little better 4= Same 5= A little worse 6= Much worse 7= Very much worse. Least squares (LS) means were calculated using mixed model repeated measures adjusting for treatment + visit + treatment*visit + age*acheifl + age + concomitant use of acetylcholinesterase inhibitor (AChEI).
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline CGIC data.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Number analyzed (Participants) | 73 | 77 | 69 | 55
Score on a scale | 4.0 (0.13) | 3.8 (0.12) | 3.3 (0.13) | 3.1 (0.15)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY3154207; Test type: Superiority; p = 0.273, Mixed Models Analysis; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.54 to 0.15]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY3154207; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.02 to -0.30]
Statistical Analysis 3: Comparison: Placebo vs 75 mg LY3154207; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.9, 95% CI 2-sided [-1.29 to -0.53]

3. Secondary Outcome: Change From Baseline on the CDR-CCB Power of Attention (PoA) Composite Score
Description: The PoA is a composite score derived from the CDR-CCB that measures the intensity of concentration (ability to focus attention): the faster the responses, the more processes are being brought to bear upon the task. Power of attention is calculated from the sum of three cognitive function speed tests: simple reaction time, choice reaction time and the speed of detections in digit vigilance task. Score ranges from 450 milliseconds - 61500 milliseconds. A low score reflects a fast reaction time and a high intensity of concentration. A positive change from baseline reflects impairment compared to the baseline assessment Values are calculated by a computer and higher scores mean better outcome. LS means were calculated using mixed model repeated measures adjusting for baseline total Score + treatment + visit + treatment*Visit + visit*baseline total Score + age + concomitant use of AChEI.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline CDR-CCB PoA data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Number analyzed (Participants) | 69 | 73 | 65 | 54
Units on a scale | 64.14 (48.681) | -6.57 (48.396) | -42.88 (49.804) | -59.58 (54.379)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY3154207; Test type: Superiority; p = 0.303, Mixed Models Analysis; Mean Difference (Net) = -70.71, 95% CI 2-sided [-205.53 to 64.11], Standard Error of Mean 68.495
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY3154207; Test type: Superiority; p = 0.125, Mixed Models Analysis; Median Difference (Net) = -107.02, 95% CI 2-sided [-244.09 to 30.06], Standard Error of Mean 69.647
Statistical Analysis 3: Comparison: Placebo vs 75 mg LY3154207; Test type: Superiority; p = 0.091, Mixed Models Analysis; Mean Difference (Net) = -123.72, 95% CI 2-sided [-267.18 to 19.74], Standard Error of Mean 72.892

4. Secondary Outcome: Change From Baseline in the 13-item Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog13)
Description: The ADAS is a rater administered instrument that was designed to assess the severity of the dysfunction in the cognitive and noncognitive behaviors characteristic of persons with AD. The cognitive subscale of the ADAS that was used as the primary efficacy measure consists of 13 items assessing areas of cognitive function most typically impaired in AD: orientation, verbal memory, language, praxis, delayed free recall, digit cancellation. The ADAS--Cog13 scale ranges from 0 to 85. Higher scores indicate greater disease severity. LS means were calculated using mixed model repeated measures adjusting for baseline total Score + treatment + visit + treatment*Visit + visit*baseline total Score + age + concomitant use of AChEI.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline ADAS-Cog13 data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Number analyzed (Participants) | 68 | 73 | 67 | 54
Units on a scale | -0.71 (0.707) | -1.11 (0.691) | -1.42 (0.720) | -1.59 (0.799)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY3154207; Test type: Superiority; p = 0.686, Mixed Models Analysis; Mean Difference (Net) = -0.40, 95% CI 2-sided [-2.34 to 1.54], Standard Error of Mean 0.985
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY3154207; Test type: Superiority; p = 0.485, Mixed Models Analysis; Mean Difference (Net) = -0.71, 95% CI 2-sided [-2.70 to 1.28], Standard Error of Mean 1.011
Statistical Analysis 3: Comparison: Placebo vs 75 mg LY3154207; Test type: Superiority; p = 0.406, Mixed Models Analysis; Mean Difference (Net) = -0.89, 95% CI 2-sided [-2.98 to 1.21], Standard Error of Mean 1.064

5. Secondary Outcome: Change From Screening in the Montreal Cognitive Assessment (MoCA) Score
Description: The Montreal Cognitive Assessment is a screening tool for global cognitive function with a total score ranging from 0 to 30 units on a scale. The MoCA is divided into 7 subscores (maximum possible subscore): visuospatial/executive (5 points), naming (3 points), memory (5 points for delayed recall), attention (6 points), language (3 points), abstraction (2 points) and orientation to time and place (6 points). A score of 26-30 is normal. A score less than 26 is considered as mild cognitive impairment. Higher values represent a better outcome. LS means were calculated using mixed model repeated measures adjusting for baseline total Score + treatment + visit + treatment*Visit + visit*baseline total Score + age + concomitant use of AChEI.
Time Frame: Screening (Baseline), Week 12
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline MoCA data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Number analyzed (Participants) | 71 | 76 | 68 | 55
Units on a scale | 0.90 (0.432) | 1.34 (0.423) | 1.12 (0.448) | 1.84 (0.496)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY3154207; Test type: Superiority; p = 0.464, Mixed Models Analysis; Mean Difference (Net) = 0.44, 95% CI 2-sided [-0.74 to 1.63], Standard Error of Mean 0.603
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY3154207; Test type: Superiority; p = 0.720, Mixed Models Analysis; Mean Difference (Net) = 0.22, 95% CI 2-sided [-1.00 to 1.45], Standard Error of Mean 0.623
Statistical Analysis 3: Comparison: Placebo vs 75 mg LY3154207; Test type: Superiority; p = 0.149, Mixed Models Analysis; Mean Difference (Net) = 0.95, 95% CI 2-sided [-0.34 to 2.24], Standard Error of Mean 0.655

6. Secondary Outcome: Change From Baseline in the Neuropsychiatric Inventory (NPI) Total Score and Individual Item Scores
Description: The NPI is a condition-specific measure designed to assess neuropsychiatric disturbances in people with Alzheimer Disease (AD),as well as other related dementing disorders.It assesses 12 behavioral disturbances,namely delusions,hallucinations,depression/dysphoria,anxiety,agitation/aggression,elation/euphoria,disinhibition,irritability/lability,apathy, aberrant motor activity, night-time behavior disturbances,and appetite/eating abnormalities.The frequency scored from 0 (never) to 4 (very frequently).The Severity scored from 0 (none) to 3 (marked).The domain score is obtained by multiplying frequency and severity scores.The total NPI score is sum total of all of individual domain scores (0-144).Higher score indiciates more abnormal behaviors.LS means were calculated using mixed model repeated measures adjusting for baseline total score + treatment + visit + treatment*visit + visit*baseline total score + age + concomitant use of AChEI.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline NPI score data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Number analyzed (Participants) | 73 | 77 | 66 | 55
Units on a scale
  Total Score: number analyzed (Participants) | 73 | 77 | 65 | 55
  Total Score | -1.62 (0.868) | -2.24 (0.852) | -3.32 (0.920) | -2.37 (1.005)
  Delusions: number analyzed (Participants) | 73 | 77 | 66 | 54
  Delusions | 0.13 (0.124) | -0.04 (0.121) | -0.25 (0.130) | 0.02 (0.144)
  Hallucinations | -0.09 (0.131) | -0.11 (0.128) | -0.44 (0.137) | -0.38 (0.151)
  Agitation/Aggression: number analyzed (Participants) | 71 | 77 | 66 | 55
  Agitation/Aggression | 0.04 (0.130) | -0.06 (0.126) | -0.02 (0.135) | -0.20 (0.148)
  Depression/Dysphoria | -0.22 (0.155) | -0.16 (0.151) | -0.33 (0.164) | -0.35 (0.179)
  Anxiety: number analyzed (Participants) | 73 | 77 | 65 | 55
  Anxiety | -0.15 (0.141) | -0.15 (0.138) | 0.07 (0.149) | -0.22 (0.163)
  Elation/Euphoria: number analyzed (Participants) | 73 | 77 | 65 | 55
  Elation/Euphoria | 0.14 (0.069) | 0.03 (0.068) | 0.00 (0.074) | 0.06 (0.080)
  Apathy/Indifference: number analyzed (Participants) | 73 | 77 | 65 | 55
  Apathy/Indifference | -0.36 (0.191) | -0.81 (0.186) | -0.68 (0.202) | -0.55 (0.220)
  Disinhibition: number analyzed (Participants) | 73 | 77 | 65 | 55
  Disinhibition | -0.13 (0.082) | -0.11 (0.080) | 0.21 (0.087) | -0.09 (0.095)
  Irritability/Lability: number analyzed (Participants) | 73 | 77 | 65 | 55
  Irritability/Lability | -0.19 (0.130) | -0.43 (0.127) | -0.25 (0.137) | 0.02 (0.150)
  Aberrant Motor Behavior: number analyzed (Participants) | 73 | 77 | 65 | 55
  Aberrant Motor Behavior | -0.13 (0.106) | 0.03 (0.103) | -0.23 (0.112) | -0.09 (0.122)
  Sleep/Nighttime Behavior Disorders | -0.19 (0.287) | 0.00 (0.278) | -0.58 (0.302) | -0.30 (0.329)
  Appetite/Eating Disorders | -0.37 (0.270) | -0.47 (0.263) | -0.80 (0.284) | -0.27 (0.311)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY3154207; Total Score; Test type: Superiority; p = 0.607, Mixed Models Analysis; Mean Difference (Net) = -0.62, 95% CI 2-sided [-3.01 to 1.76], Standard Error of Mean 1.213
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY3154207; Total Score; Test type: Superiority; p = 0.180, Mixed Models Analysis; Mean Difference (Net) = -1.70, 95% CI 2-sided [-4.19 to 0.79], Standard Error of Mean 1.265
Statistical Analysis 3: Comparison: Placebo vs 75 mg LY3154207; Total Score; Test type: Superiority; p = 0.572, Mixed Models Analysis; Mean Difference (Net) = -0.75, 95% CI 2-sided [-3.36 to 1.86], Standard Error of Mean 1.325
Statistical Analysis 4: Comparison: Placebo vs 10 mg LY3154207; Delusions; Test type: Superiority; p = 0.320, Mixed Models Analysis; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.51 to 0.17], Standard Error of Mean 0.173
Statistical Analysis 5: Comparison: Placebo vs 30 mg LY3154207; Delusions; Test type: Superiority; p = 0.037, Mixed Models Analysis; Mean Difference (Net) = -0.38, 95% CI 2-sided [-0.73 to -0.02], Standard Error of Mean 0.180
Statistical Analysis 6: Comparison: Placebo vs 75 mg LY3154207; Delusions; Test type: Superiority; p = 0.558, Mixed Models Analysis; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.49 to 0.26], Standard Error of Mean 0.190
Statistical Analysis 7: Comparison: Placebo vs 10 mg LY3154207; Hallucinations; Test type: Superiority; p = 0.924, Mixed Models Analysis; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.38 to 0.34], Standard Error of Mean 0.182
Statistical Analysis 8: Comparison: Placebo vs 30 mg LY3154207; Hallucinations; Test type: Superiority; p = 0.061, Mixed Models Analysis; Mean Difference (Net) = -0.36, 95% CI 2-sided [-0.73 to 0.02], Standard Error of Mean 0.189
Statistical Analysis 9: Comparison: Placebo vs 75 mg LY3154207; Hallucinations; Test type: Superiority; p = 0.148, Mixed Models Analysis; Mean Difference (Net) = -0.29, 95% CI 2-sided [-0.68 to 0.10], Standard Error of Mean 0.199
Statistical Analysis 10: Comparison: Placebo vs 10 mg LY3154207; Agitation/Aggression; Test type: Superiority; p = 0.552, Mixed Models Analysis; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.46 to 0.25], Standard Error of Mean 0.180
Statistical Analysis 11: Comparison: Placebo vs 30 mg LY3154207; Agitation/Aggression; Test type: Superiority; p = 0.735, Mixed Models Analysis; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.43 to 0.31], Standard Error of Mean 0.188
Statistical Analysis 12: Comparison: Placebo vs 75 mg LY3154207; Agitation/Aggression; Test type: Superiority; p = 0.224, Mixed Models Analysis; Mean Difference (Net) = -0.24, 95% CI 2-sided [-0.63 to 0.15], Standard Error of Mean 0.197
Statistical Analysis 13: Comparison: Placebo vs 10 mg LY3154207; Depression/Dysphoria; Test type: Superiority; p = 0.783, Mixed Models Analysis; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.37 to 0.48], Standard Error of Mean 0.216
Statistical Analysis 14: Comparison: Placebo vs 30 mg LY3154207; Depression/Dysphoria; Test type: Superiority; p = 0.640, Mixed Models Analysis; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.55 to 0.34], Standard Error of Mean 0.226
Statistical Analysis 15: Comparison: Placebo vs 75 mg LY3154207; Depression/Dysphoria; Test type: Superiority; p = 0.592, Mixed Models Analysis; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.59 to 0.34], Standard Error of Mean 0.236
Statistical Analysis 16: Comparison: Placebo vs 10 mg LY3154207; Anxiety; Test type: Superiority; p = 0.993, Mixed Models Analysis; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.39 to 0.39], Standard Error of Mean 0.197
Statistical Analysis 17: Comparison: Placebo vs 30 mg LY3154207; Anxiety; Test type: Superiority; p = 0.290, Mixed Models Analysis; Mean Difference (Net) = 0.22, 95% CI 2-sided [-0.19 to 0.62], Standard Error of Mean 0.205
Statistical Analysis 18: Comparison: Placebo vs 75 mg LY3154207; Anxiety; Test type: Superiority; p = 0.722, Mixed Models Analysis; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.50 to 0.35], Standard Error of Mean 0.215
Statistical Analysis 19: Comparison: Placebo vs 10 mg LY3154207; Elation/Euphoria; Test type: Superiority; p = 0.246, Mixed Models Analysis; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.30 to 0.08], Standard Error of Mean 0.097
Statistical Analysis 20: Comparison: Placebo vs 30 mg LY3154207; Elation/Euphoria; Test type: Superiority; p = 0.175, Mixed Models Analysis; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.34 to 0.06], Standard Error of Mean 0.101
Statistical Analysis 21: Comparison: Placebo vs 75 mg LY3154207; Elation/Euphoria; Test type: Superiority; p = 0.482, Mixed Models Analysis; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.28 to 0.13], Standard Error of Mean 0.106
Statistical Analysis 22: Comparison: Placebo vs 10 mg LY3154207; Apathy/Indifference; Test type: Superiority; p = 0.091, Mixed Models Analysis; Mean Difference (Net) = -0.45, 95% CI 2-sided [-0.97 to 0.07], Standard Error of Mean 0.266
Statistical Analysis 23: Comparison: Placebo vs 30 mg LY3154207; Apathy/Indifference; Test type: Superiority; p = 0.248, Mixed Models Analysis; Mean Difference (Net) = -0.32, 95% CI 2-sided [-0.87 to 0.23], Standard Error of Mean 0.278
Statistical Analysis 24: Comparison: Placebo vs 75 mg LY3154207; Apathy/Indifference; Test type: Superiority; p = 0.516, Mixed Models Analysis; Mean Difference (Net) = -0.19, 95% CI 2-sided [-0.76 to 0.38], Standard Error of Mean 0.290
Statistical Analysis 25: Comparison: Placebo vs 10 mg LY3154207; Disinhibition; Test type: Superiority; p = 0.875, Mixed Models Analysis; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.21 to 0.24], Standard Error of Mean 0.114
Statistical Analysis 26: Comparison: Placebo vs 30 mg LY3154207; Disinhibition; Test type: Superiority; p = 0.005, Mixed Models Analysis; Mean Difference (Net) = 0.34, 95% CI 2-sided [0.10 to 0.57], Standard Error of Mean 0.119
Statistical Analysis 27: Comparison: Placebo vs 75 mg LY3154207; Disinhibition; Test type: Superiority; p = 0.761, Mixed Models Analysis; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.21 to 0.28], Standard Error of Mean 0.125
Statistical Analysis 28: Comparison: Placebo vs 10 mg LY3154207; Irritability/Lability; Test type: Superiority; p = 0.183, Mixed Models Analysis; Mean Difference (Net) = -0.24, 95% CI 2-sided [-0.60 to 0.12], Standard Error of Mean 0.181
Statistical Analysis 29: Comparison: Placebo vs 30 mg LY3154207; Irritability/Lability; Test type: Superiority; p = 0.765, Mixed Models Analysis; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.43 to 0.31], Standard Error of Mean 0.189
Statistical Analysis 30: Comparison: Placebo vs 75 mg LY3154207; Irritability/Lability; Test type: Superiority; p = 0.279, Mixed Models Analysis; Mean Difference (Net) = 0.21, 95% CI 2-sided [-0.18 to 0.61], Standard Error of Mean 0.198
Statistical Analysis 31: Comparison: Placebo vs 10 mg LY3154207; Aberrant Motor Behavior; Test type: Superiority; p = 0.252, Mixed Models Analysis; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.12 to 0.46], Standard Error of Mean 0.147
Statistical Analysis 32: Comparison: Placebo vs 30 mg LY3154207; Aberrant Motor Behavior; Test type: Superiority; p = 0.526, Mixed Models Analysis; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.40 to 0.20], Standard Error of Mean 0.154
Statistical Analysis 33: Comparison: Placebo vs 75 mg LY3154207; Aberrant Motor Behavior; Test type: Superiority; p = 0.800, Mixed Models Analysis; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.28 to 0.36], Standard Error of Mean 0.161
Statistical Analysis 34: Comparison: Placebo vs 10 mg LY3154207; Sleep/Nighttime Behavior Disorders; Test type: Superiority; p = 0.623, Mixed Models Analysis; Mean Difference (Net) = 0.20, 95% CI 2-sided [-0.59 to 0.98], Standard Error of Mean 0.400
Statistical Analysis 35: Comparison: Placebo vs 30 mg LY3154207; Sleep/Nighttime Behavior Disorders; Test type: Superiority; p = 0.354, Mixed Models Analysis; Mean Difference (Net) = -0.39, 95% CI 2-sided [-1.21 to 0.44], Standard Error of Mean 0.418
Statistical Analysis 36: Comparison: Placebo vs 75 mg LY3154207; Sleep/Nighttime Behavior Disorders; Test type: Superiority; p = 0.809, Mixed Models Analysis; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.97 to 0.75], Standard Error of Mean 0.437
Statistical Analysis 37: Comparison: Placebo vs 10 mg LY3154207; Appetite/Eating Disorders; Test type: Superiority; p = 0.790, Mixed Models Analysis; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.84 to 0.64], Standard Error of Mean 0.376
Statistical Analysis 38: Comparison: Placebo vs 30 mg LY3154207; Appetite/Eating Disorders; Test type: Superiority; p = 0.280, Mixed Models Analysis; Mean Difference (Net) = -0.42, 95% CI 2-sided [-1.20 to 0.35], Standard Error of Mean 0.392
Statistical Analysis 39: Comparison: Placebo vs 75 mg LY3154207; Appetite/Eating Disorders; Test type: Superiority; p = 0.797, Mixed Models Analysis; Mean Difference (Net) = 0.11, 95% CI 2-sided [-0.70 to 0.92], Standard Error of Mean 0.412

7. Secondary Outcome: Change From Baseline in the Epworth Sleepiness Scale (ESS) Score
Description: The ESS is a self-administered questionnaire with 8 questions. Each activity is scored on a scale ranging from 0-3, with 0 = would never fall asleep, and 3 = high chance of falling asleep. The total score ranges from 0-24, with a higher number representing an increased propensity for sleepiness. LS means were calculated using mixed model repeated measures adjusting for baseline total score + treatment + visit + treatment*visit + visit*baseline total score + age + concomitant use of AChEI.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline ESS data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Number analyzed (Participants) | 73 | 77 | 67 | 55
Units on a scale | -0.33 (0.437) | -1.04 (0.426) | -1.21 (0.452) | -1.92 (0.500)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY3154207; Test type: Superiority; p = 0.247, Mixed Models Analysis; Mean Difference (Net) = -0.71, 95% CI 2-sided [-1.91 to 0.49], Standard Error of Mean 0.610
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY3154207; Test type: Superiority; p = 0.164, Mixed Models Analysis; Mean Difference (Net) = -0.88, 95% CI 2-sided [-2.12 to 0.36], Standard Error of Mean 0.631
Statistical Analysis 3: Comparison: Placebo vs 75 mg LY3154207; Test type: Superiority; p = 0.017, Mixed Models Analysis; Mean Difference (Net) = -1.59, 95% CI 2-sided [-2.90 to -0.29], Standard Error of Mean 0.663

8. Secondary Outcome: Change From Baseline in the Movement Disorder Society's Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Total Score (Sum of Parts I-III)
Description: Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) retains the four-scale structure with a reorganization of the various subscale; (Part I; 13 items) non-motor experiences of daily living, (Part II; 13) motor experiences of daily living, (Part III; 34) motor examination, and (Part IV; 6) motor complications. The scale range for MDS-UPDRS MDS-UPDRS Part I (non-motor experiences of daily living) and Part II (motor experiences of daily living) scores, total score was 0-52, with higher scores reflecting greater severity. For MDS-UPDRS Part III (motor examination) scores, the scale range for Part III Total Score was 0-132, with higher scores reflecting greater severity. LS means were calculated using mixed model repeated measures adjusting for baseline total score + treatment + visit + treatment*visit + visit*baseline total score + age + concomitant use of AChEI + levodopa equivalency dose (LED).
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline MDS-UPDRS data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Number analyzed (Participants) | 56 | 70 | 61 | 50
Units on a scale | -0.18 (2.112) | -6.58 (1.941) | -7.56 (2.084) | -10.77 (2.287)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY3154207; Test type: Superiority; p = 0.026, Mixed Models Analysis; Mean Difference (Net) = -6.41, 95% CI 2-sided [-12.04 to -0.77], Standard Error of Mean 2.860
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY3154207; Test type: Superiority; p = 0.014, Mixed Models Analysis; Mean Difference (Net) = -7.39, 95% CI 2-sided [-13.24 to -1.53], Standard Error of Mean 2.969
Statistical Analysis 3: Comparison: Placebo vs 75 mg LY3154207; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -10.60, 95% CI 2-sided [-16.72 to -4.48], Standard Error of Mean 3.104

9. Secondary Outcome: Change From Baseline in the Penn Parkinson's Daily Activities Questionnaire-15 (PDAQ-15) Total Score
Description: The PDAQ-15 is a 15-item measure of instrumental activities of daily living (IADL) that are impacted by cognitive impairment in participants with parkinson's disease dementia (PDD). The PDAQ-15 is derived from the original 50-item scale, which has demonstrated test-retest reliability, construct validity, sensitivity, and specificity to Parkinson's disease (PD) cognitive impairment and the questionnaire is completed by the caregiver. The score range is 0 to 60, with higher scores indicating better function. LS means were calculated using mixed model repeated measures adjusting for baseline total score + treatment + visit + treatment*visit + visit*baseline total score + age + concomitant use of AChEI.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline PDAQ-15 data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Number analyzed (Participants) | 73 | 77 | 67 | 55
Units on a scale | -0.32 (0.976) | 0.23 (0.961) | 2.09 (1.018) | 1.24 (1.128)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY3154207; Test type: Superiority; p = 0.683, Mixed Models Analysis; Mean Difference (Net) = 0.56, 95% CI 2-sided [-2.13 to 3.24], Standard Error of Mean 1.362
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY3154207; Test type: Superiority; p = 0.089, Mixed Models Analysis; Mean Difference (Net) = 2.41, 95% CI 2-sided [-0.37 to 5.19], Standard Error of Mean 1.413
Statistical Analysis 3: Comparison: Placebo vs 75 mg LY3154207; Test type: Superiority; p = 0.294, Mixed Models Analysis; Mean Difference (Net) = 1.56, 95% CI 2-sided [-1.37 to 4.49], Standard Error of Mean 1.489

10. Secondary Outcome: Change From Baseline in Delis-Kaplan Executive Function System (D-KEFS) Verbal Fluency Test Score
Description: The DKEFS verbal fluency category switching test measures letter fluency, category fluency, and category switching. The score is the total number of correct words generated during each of the 60-second trials within the three conditions of the test. Scales scores vary from 0 min to N/A max (no concrete maximum). Higher score = higher ability in language processing. LS means were calculated using mixed model repeated measures adjusting for baseline total score + treatment + visit + treatment*visit + visit*baseline total score + age + concomitant use of AChEI.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline D-KEFS data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Number analyzed (Participants) | 71 | 76 | 66 | 53
Units on a scale | -0.19 (0.280) | 0.44 (0.271) | 0.88 (0.292) | 0.30 (0.325)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY3154207; Test type: Superiority; p = 0.105, Mixed Models Analysis; Mean Difference (Net) = 0.63, 95% CI 2-sided [-0.13 to 1.40], Standard Error of Mean 0.389
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY3154207; Test type: Superiority; p = 0.009, Mixed Models Analysis; Mean Difference (Net) = 1.07, 95% CI 2-sided [0.27 to 1.87], Standard Error of Mean 0.406
Statistical Analysis 3: Comparison: Placebo vs 75 mg LY3154207; Test type: Superiority; p = 0.253, Mixed Models Analysis; Mean Difference (Net) = 0.49, 95% CI 2-sided [-0.35 to 1.33], Standard Error of Mean 0.428

11. Secondary Outcome: Change in MDS-UPDRS Parts II (Motor Experiences of Daily Living) and III (Motor Exam) From Baseline to Week 12
Description: Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) retains the four-scale structure with a reorganization of the various subscale; (Part I; 13 items) non-motor experiences of daily living, (Part II; 13) motor experiences of daily living, (Part III; 34) motor examination, and (Part IV; 6) motor complications. The scale range for Part II total score was 0-52, with higher scores reflecting greater severity. For MDS-UPDRS Part III (motor examination) scores, the scale range for Part III Total Score was 0-132, with higher scores reflecting greater severity. LS means were calculated using mixed model repeated measures adjusting for baseline total score + treatment + visit + treatment*visit + visit*baseline total score + age + concomitant use of AChEI + LED dose.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline MDS-UPDRS data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Number analyzed (Participants) | 75 | 77 | 69 | 54
Units on a scale
  Motor Experiences of Daily Living: number analyzed (Participants) | 73 | 77 | 69 | 53
  Motor Experiences of Daily Living | 0.28 (0.656) | -1.45 (0.649) | -2.08 (0.700) | -3.22 (0.779)
  Motor Exam: number analyzed (Participants) | 57 | 71 | 61 | 52
  Motor Exam | -0.12 (1.343) | -3.39 (1.240) | -3.40 (1.331) | -4.35 (1.434)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY3154207; Motor Experiences of Daily Living; Test type: Superiority; p = 0.061, Mixed Models Analysis; Mean Difference (Net) = -1.74, 95% CI 2-sided [-3.56 to 0.08], Standard Error of Mean 0.923
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY3154207; Motor Experiences of Daily Living; Test type: Superiority; p = 0.014, Mixed Models Analysis; Mean Difference (Net) = -2.37, 95% CI 2-sided [-4.26 to -0.47], Standard Error of Mean 0.960
Statistical Analysis 3: Comparison: Placebo vs 75 mg LY3154207; Motor Experiences of Daily Living; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -3.50, 95% CI 2-sided [-5.50 to -1.51], Standard Error of Mean 1.013
Statistical Analysis 4: Comparison: Placebo vs 10 mg LY3154207; Motor Exam; Test type: Superiority; p = 0.074, Mixed Models Analysis; Mean Difference (Net) = -3.27, 95% CI 2-sided [-6.86 to 0.32], Standard Error of Mean 1.822
Statistical Analysis 5: Comparison: Placebo vs 30 mg LY3154207; Motor Exam; Test type: Superiority; p = 0.085, Mixed Models Analysis; Mean Difference (Net) = -3.27, 95% CI 2-sided [-7.00 to 0.45], Standard Error of Mean 1.891
Statistical Analysis 6: Comparison: Placebo vs 75 mg LY3154207; Motor Exam; Test type: Superiority; p = 0.032, Mixed Models Analysis; Mean Difference (Net) = -4.23, 95% CI 2-sided [-8.09 to -0.37], Standard Error of Mean 1.959

12. Secondary Outcome: Number of Participants Who Met the Potentially Clinically Significant Vital Signs Criteria at 3 Consecutive Time Points at Visit 3
Description: Number of participants who met the potentially clinically significant vital signs criteria at 3 consecutive time points at visit 3 were reported. In the event of an unacceptable rate of participants meeting day 1 stopping rules at other doses, adjustments to doses may be made for subsequently randomized participants at the discretion of the internal assessment committee (IAC).
Time Frame: Visit 3 (Day 1 stopping rules)
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Number analyzed (Participants) | 86 | 86 | 65 | 87
Participants | 0 | 0 | 1 | 1

13. Secondary Outcome: Change From Baseline in Clinic Blood Pressure (BP) to 8 Hours Post Dose
Description: Systolic and diastolic blood pressure obtained from ambulatory blood pressure monitoring (ABPM) was evaluated. LS means were calculated using mixed model repeated measures adjusting for baseline + treatment + visit + visit*baseline + treatment*visit.
Time Frame: Baseline, 8 Hours Post Dose
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline BP data.
Measure: Least Squares Mean (Standard Error); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Number analyzed (Participants) | 81 | 82 | 79 | 85
millimeter of mercury (mmHg)
  Sitting Systolic Blood Pressure | 9.8 (1.90) | 10.1 (1.89) | 10.4 (1.92) | 19.2 (1.87)
  Sitting Diastolic Blood Pressure | 4.6 (0.99) | 4.9 (0.98) | 5.5 (1.00) | 8.1 (0.97)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY3154207; Sitting Systolic Blood Pressure; Test type: Superiority; p = 0.898, Mixed Models Analysis; Mean Difference (Net) = 0.3, 95% CI 2-sided [-4.92 to 5.61]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY3154207; Sitting Systolic Blood Pressure; Test type: Superiority; p = 0.821, Mixed Models Analysis; Mean Difference (Net) = 0.6, 95% CI 2-sided [-4.71 to 5.94]
Statistical Analysis 3: Comparison: Placebo vs 75 mg LY3154207; Sitting Systolic Blood Pressure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 9.4, 95% CI 2-sided [4.11 to 14.61]
Statistical Analysis 4: Comparison: Placebo vs 10 mg LY3154207; Sitting Diastolic Blood Pressure; Test type: Superiority; p = 0.805, Mixed Models Analysis; Mean Difference (Net) = 0.3, 95% CI 2-sided [-2.40 to 3.08]
Statistical Analysis 5: Comparison: Placebo vs 30 mg LY3154207; Sitting Diastolic Blood Pressure; Test type: Superiority; p = 0.513, Mixed Models Analysis; Mean Difference (Net) = 0.9, 95% CI 2-sided [-1.85 to 3.69]
Statistical Analysis 6: Comparison: Placebo vs 75 mg LY3154207; Sitting Diastolic Blood Pressure; Test type: Superiority; p = 0.011, Mixed Models Analysis; Mean Difference (Net) = 3.6, 95% CI 2-sided [0.83 to 6.28]

14. Secondary Outcome: Change From Baseline in Pulse Rate to 8 Hours Post Dose
Description: Pulse rate obtained from ABPM was evaluated. Pulse rate measurements will occur at time 0 and every 60 minutes thereafter up to 8 hours and pulse rate measurements will be done in the seated position only. LS means were calculated using mixed model repeated measures adjusting for baseline + treatment + visit + visit*baseline + treatment*visit.
Time Frame: Baseline, 8 Hours Post Dose
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline pulse rate data.
Measure: Least Squares Mean (Standard Error); unit: beats/min
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Number analyzed (Participants) | 81 | 82 | 79 | 85
beats/min | -2.2 (0.94) | 0.2 (0.95) | 1.3 (0.95) | 6.4 (0.93)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY3154207; Test type: Superiority; p = 0.065, Mixed Models Analysis; Mean Difference (Net) = 2.5, 95% CI 2-sided [-0.16 to 5.08]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY3154207; Test type: Superiority; p = 0.008, Mixed Models Analysis; Mean Difference (Net) = 3.6, 95% CI 2-sided [0.93 to 6.21]
Statistical Analysis 3: Comparison: Placebo vs 75 mg LY3154207; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 8.7, 95% CI 2-sided [6.06 to 11.27]

15. Secondary Outcome: Change From Baseline In-clinic BP to Week 12
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) obtained from ambulatory blood pressure monitoring (ABPM) was evaluated. LS means were calculated using mixed model repeated measures adjusting for baseline + treatment + visit + visit*baseline + treatment*visit.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline BP data.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Number analyzed (Participants) | 74 | 77 | 65 | 56
millimeters of mercury (mmHg)
  Sitting Systolic Blood Pressure | -1.2 (1.22) | 0.5 (1.19) | 0.1 (1.29) | 3.0 (1.38)
  Sitting Diastolic Blood Pressure | -0.9 (0.71) | -1.0 (0.70) | -0.2 (0.75) | 0.3 (0.80)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY3154207; Sitting Systolic Blood Pressure; Test type: Superiority; p = 0.339, Mixed Models Analysis; Mean Difference (Net) = 1.6, 95% CI 2-sided [-1.72 to 4.99]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY3154207; Sitting Systolic Blood Pressure; Test type: Superiority; p = 0.486, Mixed Models Analysis; Mean Difference (Net) = 1.2, 95% CI 2-sided [-2.26 to 4.73]
Statistical Analysis 3: Comparison: Placebo vs 75 mg LY3154207; Sitting Systolic Blood Pressure; Test type: Superiority; p = 0.024, Mixed Models Analysis; Mean Difference (Net) = 4.2, 95% CI 2-sided [0.56 to 7.81]
Statistical Analysis 4: Comparison: Placebo vs 10 mg LY3154207; Sitting Diastolic Blood Pressure; Test type: Superiority; p = 0.935, Mixed Models Analysis; Mean Difference (Net) = -0.1, 95% CI 2-sided [-2.04 to 1.88]
Statistical Analysis 5: Comparison: Placebo vs 30 mg LY3154207; Sitting Diastolic Blood Pressure; Test type: Superiority; p = 0.505, Mixed Models Analysis; Mean Difference (Net) = 0.7, 95% CI 2-sided [-1.34 to 2.72]
Statistical Analysis 6: Comparison: Placebo vs 75 mg LY3154207; Sitting Diastolic Blood Pressure; Test type: Superiority; p = 0.266, Mixed Models Analysis; Mean Difference (Net) = 1.22, 95% CI 2-sided [-0.91 to 3.30]

16. Secondary Outcome: Change From Baseline in Pulse Rate to Week 12
Description: as for outcome 14
Time Frame: Baseline, Week 12
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: beats/min
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Number analyzed (Participants) | 74 | 77 | 65 | 56
beats/min | -0.2 (0.67) | 0.3 (0.66) | 1.5 (0.71) | 2.6 (0.75)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY3154207; Test type: Superiority; p = 0.550, Mixed Models Analysis; Mean Difference (Net) = 0.6, 95% CI 2-sided [-1.28 to 2.41]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY3154207; Test type: Superiority; p = 0.069, Mixed Models Analysis; Mean Difference (Net) = 1.8, 95% CI 2-sided [-0.14 to 3.68]
Statistical Analysis 3: Comparison: Placebo vs 75 mg LY3154207; Test type: Superiority; p = 0.005, Mixed Models Analysis; Mean Difference (Net) = 2.9, 95% CI 2-sided [0.89 to 4.83]

17. Secondary Outcome: Change in Home Blood Pressure Measurement (HBPM), for SBP, DBP From Baseline to Week 12
Description: Systolic and diastolic blood pressure obtained from ABPM was evaluated. Participants followed a standardized measurement protocol for home blood pressure measurement, involving three consecutive measurements, taken one minute apart after a five-minute seated resting period. LS means were calculated using mixed model repeated measures adjusting for baseline + treatment + visit + visit*baseline + treatment*visit.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline BP data.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Number analyzed (Participants) | 48 | 51 | 41 | 41
mmHg
  Sitting Systolic Blood Pressure | -1.1 (2.52) | -8.2 (2.40) | 2.0 (2.58) | -2.2 (2.62)
  Sitting Diastolic Blood Pressure | 1.5 (1.50) | -2.8 (1.45) | 1.0 (1.55) | -0.8 (1.58)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY3154207; Sitting Systolic Blood Pressure; Test type: Superiority; p = 0.045, Mixed Models Analysis; Mean Difference (Net) = -7.0, 95% CI 2-sided [-13.92 to -0.15]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY3154207; Sitting Systolic Blood Pressure; Test type: Superiority; p = 0.390, Mixed Models Analysis; Mean Difference (Net) = 3.1, 95% CI 2-sided [-4.05 to 10.32]
Statistical Analysis 3: Comparison: Placebo vs 75 mg LY3154207; Sitting Systolic Blood Pressure; Test type: Superiority; p = 0.768, Mixed Models Analysis; Mean Difference (Net) = -1.1, 95% CI 2-sided [-8.32 to 6.16]
Statistical Analysis 4: Comparison: Placebo vs 10 mg LY3154207; Sitting Diastolic Blood Pressure; Test type: Superiority; p = 0.041, Mixed Models Analysis; Mean Difference (Net) = -4.3, 95% CI 2-sided [-8.48 to -0.17]
Statistical Analysis 5: Comparison: Placebo vs 30 mg LY3154207; Sitting Diastolic Blood Pressure; Test type: Superiority; p = 0.802, Mixed Models Analysis; Mean Difference (Net) = -0.5, 95% CI 2-sided [-4.81 to 3.72]
Statistical Analysis 6: Comparison: Placebo vs 75 mg LY3154207; Sitting Diastolic Blood Pressure; Test type: Superiority; p = 0.284, Mixed Models Analysis; Mean Difference (Net) = -2.4, 95% CI 2-sided [-6.67 to 1.97]

18. Secondary Outcome: Change in HBPM for Pulse Rate From Baseline to Week 12
Description: Pulse rate obtained from ABPM was evaluated. Pulse rate measurements will occur at time 0 and every 60 minutes thereafter up to week 12 and pulse rate measurements will be done in the seated position only. LS means were calculated using mixed model repeated measures adjusting for baseline + treatment + visit + visit*baseline + treatment*visit.
Time Frame: Baseline, Week 12
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: beats/min
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Number analyzed (Participants) | 48 | 51 | 41 | 41
beats/min | 1.4 (1.52) | 1.4 (1.47) | 0.7 (1.59) | 0.8 (1.62)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY3154207; Test type: Superiority; p = 0.996, Mixed Models Analysis; Mean Difference (Net) = 0.0, 95% CI 2-sided [-4.17 to 4.19]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY3154207; Test type: Superiority; p = 0.767, Mixed Models Analysis; Mean Difference (Net) = -0.7, 95% CI 2-sided [-4.99 to 3.69]
Statistical Analysis 3: Comparison: Placebo vs 75 mg LY3154207; Test type: Superiority; p = 0.791, Mixed Models Analysis; Mean Difference (Net) = -0.6, 95% CI 2-sided [-4.96 to 3.79]

19. Secondary Outcome: Change From Baseline in the Physician Withdrawal Checklist (PWC)-20 Total Score From Week 12 to In-Clinic Follow-up Visit
Description: The Penn PWC-20 is a 20-item checklist originally developed to assess the severity of withdrawal symptoms in anxiolytic medication discontinuation. To determine a change in the Intensity of Discontinuation symptoms, the PWC-20 administered by a trained clinician/rater to assess the intensity of discontinuation symptoms. The assessment has 20 items evaluated to detect withdrawal symptoms. Symptoms are rated on a scale of 0-3.
  0. Not present
  1. Mild
  2. Moderate
  3. Severe Total scores range from 0 to 60 with higher scores indicating more severe symptoms.Least squares (LS) means were calculated using mixed model analysis of covariance (ANCOVA) adjusting for predose, sequence, period, day, time, treatment, and treatment*time as fixed effects and participant within sequence and treatment as random effect.
Time Frame: Week 12, Follow-up (2 Weeks after Week 12)
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline PWC-20 data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Number analyzed (Participants) | 35 | 33 | 32 | 24
Units on a scale
  Week 12 | -1.51 (0.670) | -0.53 (0.690) | -0.47 (0.701) | 0.05 (0.811)
  Follow-up | -1.27 (0.844) | 0.12 (0.877) | 0.13 (0.904) | 3.32 (1.040)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY3154207; Week 12; Test type: Superiority; p = 0.312, ANCOVA; Mean Difference (Net) = 0.98, 95% CI 2-sided [-0.93 to 2.88]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY3154207; Week 12; Test type: Superiority; p = 0.289, ANCOVA; Mean Difference (Net) = 1.03, 95% CI 2-sided [-0.89 to 2.95]
Statistical Analysis 3: Comparison: Placebo vs 75 mg LY3154207; Week 12; Test type: Superiority; p = 0.141, ANCOVA; Mean Difference (Net) = 1.56, 95% CI 2-sided [-0.53 to 3.65]
Statistical Analysis 4: Comparison: 10 mg LY3154207 vs 30 mg LY3154207; Week 12; Test type: Superiority; p = 0.954, ANCOVA; Mean Difference (Net) = 0.06, 95% CI 2-sided [-1.89 to 2.01]
Statistical Analysis 5: Comparison: 10 mg LY3154207 vs 75 mg LY3154207; Test type: Superiority; p = 0.584, ANCOVA; Mean Difference (Net) = 0.59, 95% CI 2-sided [-1.53 to 2.70]
Statistical Analysis 6: Comparison: 30 mg LY3154207 vs 75 mg LY3154207; Week 12; Test type: Superiority; p = 0.623, ANCOVA; Mean Difference (Net) = 0.53, 95% CI 2-sided [-1.59 to 2.65]
Statistical Analysis 7: Comparison: Placebo vs 10 mg LY3154207; Follow-up; Test type: Superiority; p = 0.256, ANCOVA; Mean Difference (Net) = 1.39, 95% CI 2-sided [-1.02 to 3.79]
Statistical Analysis 8: Comparison: Placebo vs 30 mg LY3154207; Follow-up; Test type: Superiority; p = 0.258, ANCOVA; Mean Difference (Net) = 1.41, 95% CI 2-sided [-1.04 to 3.86]
Statistical Analysis 9: Comparison: Placebo vs 75 mg LY3154207; Follow-up; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 4.59, 95% CI 2-sided [1.93 to 7.25]
Statistical Analysis 10: Comparison: 10 mg LY3154207 vs 30 mg LY3154207; Follow-up; Test type: Superiority; p = 0.988, ANCOVA; Mean Difference (Net) = 0.02, 95% CI 2-sided [-2.47 to 2.51]
Statistical Analysis 11: Comparison: 10 mg LY3154207 vs 75 mg LY3154207; Follow-up; Test type: Superiority; p = 0.020, ANCOVA; Mean Difference (Net) = 3.20, 95% CI 2-sided [0.51 to 5.90]
Statistical Analysis 12: Comparison: 30 mg LY3154207 vs 75 mg LY3154207; Follow-up; Test type: Superiority; p = 0.022, ANCOVA; Mean Difference (Net) = 3.18, 95% CI 2-sided [0.46 to 5.91]

20. Secondary Outcome: Pharmacokinetics (PK): Steady-State Trough Plasma Concentrations of LY3154207
Description: Trough measurements of LY3154207 concentration in plasma at Day 1, Day 7, Day 14, Day 42 and Day 84 was evaluated.
Time Frame: Day 1: 1-3 hours post-dose; Day 7, Day 14 and Day 42: post-dose; Day 84: pre-dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
Number analyzed (Participants) | 86 | 77 | 81
nanogram per milliliter (ng/mL)
  Day 1 | 34.95 (28.82) | 89.36 (88.03) | 223.30 (208.63)
  Day 7: number analyzed (Participants) | 80 | 77 | 70
  Day 7 | 50.53 (38.20) | 123.61 (100.89) | 297.35 (242.47)
  Day 14: number analyzed (Participants) | 81 | 71 | 69
  Day 14 | 45.85 (33.61) | 129.24 (89.24) | 321.65 (253.11)
  Day 42: number analyzed (Participants) | 74 | 66 | 61
  Day 42 | 44.25 (33.93) | 149.22 (122.01) | 333.40 (257.74)
  Day 84: number analyzed (Participants) | 68 | 63 | 56
  Day 84 | 25.01 (30.43) | 59.39 (58.20) | 126.53 (197.67)

ADVERSE EVENTS:
Time Frame: Up To 4 Months
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Placebo | 10 mg LY3154207 | 30 mg LY3154207 | 75 mg LY3154207
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/86 | 1/85 | 1/87
Serious Adverse Events (participants affected / at risk) | 3/86 | 5/86 | 3/85 | 10/87
Other Adverse Events (participants affected / at risk) | 20/86 | 26/86 | 30/85 | 43/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=86) | 10 mg LY3154207 (N=86) | 30 mg LY3154207 (N=85) | 75 mg LY3154207 (N=87)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster meningoencephalitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemianaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=86) | 10 mg LY3154207 (N=86) | 30 mg LY3154207 (N=85) | 75 mg LY3154207 (N=87)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 5 (7) | 2 (4)
Nausea (Gastrointestinal disorders) | 3 (5) | 2 (2) | 7 (8) | 8 (9)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2) | 7 (8)
Fatigue (General disorders) | 4 (4) | 2 (2) | 1 (1) | 9 (9)
Urinary tract infection (Infections and infestations) | 2 (2) | 5 (5) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (10) | 12 (17) | 6 (7) | 12 (16)
Dizziness (Nervous system disorders) | 4 (4) | 4 (4) | 6 (6) | 9 (10)
Dyskinesia (Nervous system disorders) | 2 (2) | 2 (2) | 3 (3) | 5 (6)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 8 (8) | 7 (8)
Hallucination (Psychiatric disorders) | 4 (4) | 2 (2) | 5 (5) | 9 (9)
Insomnia (Psychiatric disorders) | 0 (0) | 4 (4) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/09/NCT03305809/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT03305809/SAP_001.pdf